CLINICAL TRIAL: NCT05682521
Title: Scoliosis and Postural Deformity Evaluation in Famagusta Region Secondary Schools
Status: Completed | Type: Observational
Sponsor: Eastern Mediterranean University (Other)
Responsible Party: Principal Investigator, Tuğba Paksoy, Physiotherapist, Eastern Mediterranean University
Other Study IDs: ETK00-2022-0220
Record Dates: First submitted 2022-12-25; First posted 2023-01-12 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2023-09

CONDITIONS: Scoliosis Idiopathic Adolescent
Keywords: Scoliosis Idiopathic Adolescent; School screening; Prevalence; Scoliometer; Adams test

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of the study is to evaluate scoliosis and postural deformities in secondary school students in Famagusta region. Secondary school students who meet the inclusion criteria will be included in the study, which will be conducted in the form of screening in public and private schools in the Famagusta region of the Turkish Republic of Northern Cyprus. Sociodemographic information of the individuals will be obtained first. Then, Adam's forward bending test, trunk rotation angle with scoliometer, foot posture index and New York posture index will be evaluated. Evaluations will be made within a single day.

DETAILED DESCRIPTION:
The term scoliosis originates from the ancient Greek word "scolios" (curvature) and was first used by Galen around AD 130-201. Scoliosis is a common three-dimensional deformity that causes severe postural impairment in advanced stages. It is generally defined as a curvature of the spine towards lateral flexion in the frontal plane and towards rotation in the transverse plane. Scoliosis is divided into idiopathic and non-idiopathic. Although the etiology of idiopathic scoliosis is not known exactly, it is thought that secondary causes such as genetic, hormonal and biomechanical factors and neuromuscular problems contribute to the development of scoliosis. Scoliosis; It is divided into different classes according to the age of onset, etiology, type and severity of the curvature. The most common type of scoliosis in the community is Adolescent Idiopathic Scoliosis (AIS). The Scoliosis Research Society defines adolescent idiopathic scoliosis (AIS) as a curve of Cobb angle ≥10°.

The incidence of adolescent idiopathic scoliosis (AIS) in healthy children is 2 - 4%. In Turkey, the prevalence of AIS has been reported as 2.3% in children aged 10-15 years. AIS begins in early puberty. The prevalence and severity of curvature are higher in girls than boys. While the prevalence of AIS aged 10-15 years in Turkey is 3.07% in girls, it is 1.49% in boys. Likewise, women are 8 times more prone to development of prognosis in curvature than men.

School screenings in scoliosis are very important in terms of early diagnosis, prevention or protection of deformity progression without surgical intervention. Scoliosis Research Society states that it is appropriate to perform annual routine screenings at the age of 10-14 years. Studies have been carried out in terms of early diagnosis of scoliosis worldwide and the importance of school screening as an early diagnosis method has been emphasized. According to recent literature studies, the prevalence of Adolescent Idiopathic Scoliosis (AIS) in school surveys has been shown within wide limits such as 0.47%-5.2%.

The aim of this study is that many school screening studies for scoliosis have been conducted in the literature both in the world and in Turkey, but there is no scoliosis and postural disorder screening data in TRNC. It is aimed to create an epidemiological database by calculating the prevalence of scoliosis in the 10-15 age group in secondary schools in the Famagusta region of the Turkish Republic of Northern Cyprus, as well as to evaluate postural deformities. It is expected that the data obtained will increase awareness about the incidence of scoliosis and contribute to the early diagnosis and treatment of curvature. Thus, in the long term, the development of severe spinal deformities and the medical problems caused by these deformities will be prevented.

Research Questions:

Research question 1: What is the incidence of scoliosis in secondary school students in Famagusta? Research question 2. What is the incidence of postural deformity in secondary school students in Famagusta?

Material and Method:

Secondary school students who meet the inclusion criteria will be included in the study, which will be conducted in the form of screening in public and private schools in the Famagusta region of the Turkish Republic of Northern Cyprus. Sociodemographic information of the individuals will be obtained first. Then, Adam's forward bending test, trunk rotation angle with scoliometer, foot posture index and New York posture index will be evaluated. Evaluations will be made within a single day. The sample size of the study was calculated using Epi InfoTM version 7. The initial sample size was calculated as 386 people in order to make an estimation in the 95% confidence interval under the assumptions that the population size of the study would be 2500, the expected prevalence rate would be 5%, the margin of error +/- 2%, and the pattern effect would be 1. Considering that there may be those who did not accept to participate in the study, this sample size was increased by 20% and the final sample size was calculated as 463 people.

Evaluations to be applied to the Subject:

Socio-demographic Form: In the first evaluation, socio-demographic informationof subjects such as age, height, body weight will be obtained through a form.

Adam's Forward Bend Test: This test is also known as the forward bend test. The test will be applied in a way that the boys are completely naked on the top and the girls are only athletes. With the shoes taken off, the feet together and the knee extended, the children will be asked to bend forward with their hips at a 90 degree angle, the arms will swing down freely and the palms will be facing each other. In case of scoliosis, it will be checked whether there is a rotational protrusion or asymmetry in the back as a result of the deformity of the spine in the ribs.

Body Rotation Angle Assessment: The person measuring with the scoliometer should sit in a chair behind the person to be evaluated. The person to be examined should keep his arms at head level and lean forward until the shoulders and hips are at the same level, and in this position, deviations in the scoliometer will be checked in the thoracic (T7 level), thoracolumbar (T12 level) and lumbar (L3 level) regions. Studies have shown that 7° deviation in the scoliometer corresponds to approximately 20° in the scoliosis Cobb angle of the spine. In the evaluations, students with scoliometer measurements of 7° and above will be informed about the suspicion of scoliosis and directed to the physician.

New York Posture Assessment Scale: In this evaluation system, postural changes that may occur in 13 different parts of the body are scored observationally.

Evaluation of Foot Postures: Foot posture will be assessed by the Foot PostureIndex (FPI).

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 10 - 15
* Volunteering to participate in the study
* Not having neuromuscular scoliosis

Ages: 10 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Students between the ages of 10-15 studying at secondary schools in the Famagusta region will be included in the study.
Sampling Method: Probability Sample
Enrollment: 440 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
Body Rotation Angle Evaluation with Scoliometer | 9 months
  The individual is asked to bend forward 90 degrees by joining his hands together. Measurements will be made from the thoracic, thoracalumbar and lumbar regions with a scoliometer.

SECONDARY OUTCOMES:
Adam's Forward Bend Test | 9 months
  Boys will be tested completely naked on top, and girls will be only athletes. With the shoes taken off, the feet together and the knee extended, the children will be asked to bend forward with their hips at a 90 degree angle, the arms will swing down freely and the palms will be facing each other. In case of scoliosis, it will be checked whether there is a rotational protrusion or asymmetry in the back as a result of the deformity of the spine in the ribs.
New York Posture Rating Scale | 9 months
  In this evaluation system, postural changes that may occur in 13 different parts of the body are scored observationally. Accordingly, five (5) points are given if the person's posture is correct, three (3) points if moderately impaired, and one (1) point if severely impaired. The total score obtained as a result of the test is a maximum of 65 and a minimum of 13. Standard evaluation criteria developed for this test are defined as "very good" if the total score is ≥45, "good" if 40-44, "moderate" if 30-39, "poor" if 20-29, and "poor" if it is ≤19.
Foot Posture Index | 9 months
  During the evaluation, individuals will be asked to stand still and in a relaxed position. The scale has 6 subheadings. The value of each question varies between -2 and +2 points. - values show supination, that is, increased MLA height, while + values show pronation, that is, decreased MLA height. As a result of the scale, the scores that individuals can get vary between -12 and +12. The six subheadings of the scale are palpation of the talus head, upper and lower slope of the lateral malleolus, calcaneal inversion-eversion, joint protrusion in the talonavicular region, MLA compliance, and forefoot abduction/adduction.

CONTACTS AND LOCATIONS:
Overall Officials: Tuğba PAKSOY, Bachelor, Principal Investigator — Eastern Mediterranean University; Yasin YURT, Associate professor, Study Director — Eastern Mediterranean University
Locations (1):
- Eastern Mediterranean University, Faculty of Health Sciences, Physiotherapy and Rehabilitation Department, Mersin, Famagusta, Turkey (Türkiye)

REFERENCES:
- [Background] Konieczny MR, Senyurt H, Krauspe R. Epidemiology of adolescent idiopathic scoliosis. J Child Orthop. 2013 Feb;7(1):3-9. doi: 10.1007/s11832-012-0457-4. Epub 2012 Dec 11. PMID 24432052
- [Background] Weinstein SL, Dolan LA, Cheng JC, Danielsson A, Morcuende JA. Adolescent idiopathic scoliosis. Lancet. 2008 May 3;371(9623):1527-37. doi: 10.1016/S0140-6736(08)60658-3. PMID 18456103
- [Background] Yaman O, Dalbayrak S. Idiopathic scoliosis. Turk Neurosurg. 2014;24(5):646-57. doi: 10.5137/1019-5149.JTN.8838-13.0. PMID 25269032
- [Background] Burwell RG, James NJ, Johnson F, Webb JK, Wilson YG. Standardised trunk asymmetry scores. A study of back contour in healthy school children. J Bone Joint Surg Br. 1983 Aug;65(4):452-63. doi: 10.1302/0301-620X.65B4.6874719.
- [Background] Brooks HL, Azen SP, Gerberg E, Brooks R, Chan L. Scoliosis: A prospective epidemiological study. J Bone Joint Surg Am. 1975 Oct;57(7):968-72. PMID 1194304
- [Background] Jada A, Mackel CE, Hwang SW, Samdani AF, Stephen JH, Bennett JT, Baaj AA. Evaluation and management of adolescent idiopathic scoliosis: a review. Neurosurg Focus. 2017 Oct;43(4):E2. doi: 10.3171/2017.7.FOCUS17297. PMID 28965447
- [Background] Cheng JC, Castelein RM, Chu WC, Danielsson AJ, Dobbs MB, Grivas TB, Gurnett CA, Luk KD, Moreau A, Newton PO, Stokes IA, Weinstein SL, Burwell RG. Adolescent idiopathic scoliosis. Nat Rev Dis Primers. 2015 Sep 24;1:15030. doi: 10.1038/nrdp.2015.30. PMID 27188385
- [Background] Picault C, deMauroy JC, Mouilleseaux B, Diana G. Natural history of idiopathic scoliosis in girls and boys. Spine (Phila Pa 1976). 1986 Oct;11(8):777-8. doi: 10.1097/00007632-198610000-00004. No abstract available. PMID 3810291
- [Background] De Wilde L, Plasschaert F, Cattoir H, Uyttendaele D. Examination of the back using the Bunnell scoliometer in a Belgian school population around puberty. Acta Orthop Belg. 1998 Jun;64(2):136-43. PMID 9689752
- [Background] Redmond AC, Crosbie J, Ouvrier RA. Development and validation of a novel rating system for scoring standing foot posture: the Foot Posture Index. Clin Biomech (Bristol). 2006 Jan;21(1):89-98. doi: 10.1016/j.clinbiomech.2005.08.002. Epub 2005 Sep 21. PMID 16182419
- See also: 1 — https://doi.org/10.7197/cmj.v36i3.5000038449
- See also: 2 — http://turkishneurosurgery.org.tr/pdf.php?&id=1282
- See also: 4 — https://www.srs.org/professionals/online-education-and-resources/glossary/revised-glossary-of-terms
- See also: 5 — https://www.tuseb.gov.tr/enstitu/tacese/yuklemeler/adolesan/t_a_idiyopatik_skolyoz_sonucraporu.pdf
- See also: 7 — http://www.p12.nysed.gov/sss/schoolhealth/schoolhealthservices/
- See also: 8 — https://dergipark.org.tr/en/pub/jetr/issue/41952/505544